CLINICAL TRIAL: NCT03328260
Title: Prospective, Muti-institute, Single Arm, Confirmative Trial Evaluating Efficacy and Safety of High Intensity Focused Ultrasound Device (RODIN) in Women With Symptomatic Uterine Leiomyoma
Brief Title: High Intensity Focused Ultrasound in Uterine Myoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: ALPINION Medical Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APM-05
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: HIFU

INTERVENTIONS:
Device: HIFU — Transvaginal high intensity focused ultrasound to ablate uterine myoma

SUMMARY:
Aim to evaluate the efficacy of safety of newly developed, high intensity focused ultrasound device in women with symptomatic uterine leiomyoma

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal (FSH < 40 IU/L)
* Symptomatic uterine fibroids
* Willing to contracept during study period

Exclusion Criteria:

* Pregnant or willing to be pregnant in future
* Cancer in female reproductive organ is suspected or diagnosed
* Inflammation in female reproductive organ
* Poorly controlled systemic disease
* Hematocrit < 25%
* Glomerular filtration rate(GFR) <= 30ml/min
* Cannot tolerate contrast-enhanced MR or Contrast-enhanced ultrasound(CEUS)
* Cannot lie down
* Previous treatment for leiomyoma, any of ① myolysis, ② myomectomy within 1 year, ③ hormonal therapy longer than 7 days within 4 weeks
* Cannot count the number or measure volume of leiomyoma using MRI
* Leiomyomas are inadequate (location, volume, number) for intervention
* Diameter of leiomyoma is over 5 cm
* Leiomyoma is not enhanced
* Lactating women
* Cannot communicate properly
* Participating or have participated in other trials within 30 days

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Non perfused volume | treatment day
  Non perfused volume in myoma immediately after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyenggi DO, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Kim K, Hwang SI, Lee M, Son K, Kim D, Kim S, Kim YB. Efficacy and safety of transvaginal high-intensity focused ultrasound therapy in women with symptomatic uterine leiomyomas: A clinical trial. Eur J Obstet Gynecol Reprod Biol. 2021 Jan;256:302-307. doi: 10.1016/j.ejogrb.2020.11.049. Epub 2020 Nov 17. PMID 33259999